CLINICAL TRIAL: NCT02544061
Title: A Phase IIa Open-label, Randomized Study to Compare the Safety, Tolerability and Pharmacokinetics (PK) of NM-IL-12 (rHuIL-12) to Standard of Care in Subjects With Open Surgical Wounds Following Colostomy Takedown
Brief Title: NM-IL-12 (rHuIL-12) in Subjects With Open Surgical Wounds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neumedicines Inc. (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-SWI-004; W81XWH-15-2-009 (Other Grant/Funding Number: USA MED RESEARCH ACQ ACTIVITY)
Record Dates: First submitted 2015-09-03; First posted 2015-09-09 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Colostomy Stoma
Keywords: NM-IL-12, HemaMax, Safety, Stoma Takedown, Wound closure
MeSH Terms: interventions — Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NM-IL-12 plus Standard of Care (SOC) (Experimental): Single 12 µg unit subcutaneous dose of NM-IL-12 plus SOC.
  Standard wound management: wet to dry dressing care and perioperative antimicrobial therapy
  Interventions: Biological: NM-IL-12
- Placebo plus SOC (Placebo Comparator): Single subcutaneous dose of placebo plus SOC
  Standard wound management: wet to dry dressing care and perioperative antimicrobial therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: NM-IL-12 — single 12 µg unit subcutaneous (SC) dose of NM-IL-12
  Other Names: rHu-IL12, HemaMax
  Arms: NM-IL-12 plus Standard of Care (SOC)
Drug: Placebo — single subcutaneous dose
  Arms: Placebo plus SOC

SUMMARY:
The purpose of this study is to determine the safety and tolerability of NM-IL-12 relative to standard of care (SOC; control) in subjects with open surgical wounds.

DETAILED DESCRIPTION:
This is a phase IIa open-label, randomized study to compare the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of NM-IL-12 (rHuIL-12) to standard of care in subjects with open surgical wounds following colostomy takedown allowed to heal by secondary intention.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo colostomy reversal where the midline wound is closed and the stoma site (wound) is kept open to heal by secondary intention at the time of operation but expected to close between 4 and 6 weeks (per the judgment of the investigator).
* Able to receive the dose of study drug within 24-36 hours post-operatively and demonstrate stable vital signs without unresolved major organ failure/dysfunction requiring critical care/monitoring for at least 24 hours prior to receiving study drug.
* Agree to use accepted highly effective methods of birth control (defined as one that results in a low failure rate (i.e., <1% per year when used consistently and correctly) and continue for 3 months following receipt of study drug:

  1. Sexual abstinence (males and females),
  2. Vasectomized partner (females),
  3. Condom with spermicide (males) in combination with another non-hormonal barrier method (females
  4. Females on hormonal birth control should be on these medications for at least 3 years without complications.
* Agree to use accepted highly effective methods of birth control (defined as one that results in a low failure rate (i.e., <1% per year when used consistently and correctly):

  1. Sexual abstinence (males and females),Vasectomized partner (females),
  2. Condom with spermicide (males) in combination with another non-hormonal barrier method (females), must agree to use for at least 3 months following receiving the study drug.
  3. Females on hormonal birth control should be on these medications for at least 3 years without complications.
* Surgically sterile (does not have a uterus or has had bilateral tubal ligation) or post-menopausal (no menstrual period for a minimum of 1 year) (females).
* A negative serum pregnancy test at the time of enrollment into the study for women of childbearing potential.
* Laboratory values for white blood cells (WBCs), neutrophils, lymphocytes and platelets prior to study drug administration on Day 1 as shown below:

  1. WBCs > 3500 cells/µL,
  2. Neutrophils > 2000 cells/µL,
  3. Lymphocytes > 1000 cells/µL,
  4. Platelets > 140,000 /µL.
* All other clinical chemistry and coagulation laboratory values at enrollment must be either within the reference range or considered to be not clinically significant by the investigator and sponsor. Hematological laboratory values that are outside of the reference range must be reported to be above the upper limit of normal and not be reported as clinically significant.

Exclusion Criteria:

* Concurrent infections of unremovable prosthetic materials (e.g., permanent cardiac pacemaker battery packs, or joint replacement prostheses).
* Undergoing a significant major planned concomitant surgical procedure other than hysterectomy or receiving antibiotic therapy within the week (7 days) prior to the date of surgery other than perioperative antibiotic therapy.
* Preoperative evaluation that suggests an intra-abdominal process that might preclude full closure of the skin by secondary intention.
* Treatment (e.g., chemotherapy, radiation) for cancer in the last 3 months.
* Concomitant use of systemic steroid hormones, i.e. > 10 mg/day prednisone or equivalent.
* Concomitant use of any immunosuppressive or immunomodulatory drugs.
* History of Crohn's disease or Ulcerative colitis.
* Known history of drug or alcohol abuse within the past year. A positive screening urine toxicology will also exclude patients from this study.
* Medical, social or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures.
* Preoperative prothrombin time (PT), ALT, AST, and creatinine > 1.5 times upper limit of normal.
* Lactating females.
* Postsurgical life expectancy ≤ 60 days, in the investigator or sponsor's opinion.
* Refusal to accept medically indicated blood products.
* Participation within 30 days before the start (dosing) of this study in any experimental drug or device study, or currently participating in a study in which the administration of investigational drug or device within 60 days is anticipated.
* Presence of prosthetic cardiac valve.
* Known medical history (carrier or disease) of human immunodeficiency virus (HIV), Hepatitis A, Hepatitis B, or Hepatitis C, or other diseases known to be autoimmune in origin.
* Known medical history of tuberculosis or liver cirrhosis.
* Current or prior treatment with growth factors or hyperbaric therapy in the last 30 days preceding study day 1.
* History of sensitivity to the study medication, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or medical/research monitor, contraindicates their participation.
* Uncontrolled intercurrent illness, including, but not limited to, ongoing or serious active infection (not including eligible surgical wounds), symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, metastatic cancer, chronic obstructive pulmonary disease (COPD; (using home oxygen therapy).
* Insulin-requiring diabetes.
* BMI > 40.
* Any other condition that, in the opinion of the investigator, would confound or interfere with evaluation of safety of the study drug, or prevent compliance with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of NM-IL-12 (Number of subjects with adverse events) | 42 Days
  Number of subjects with adverse events as a measure of safety and tolerability

SECONDARY OUTCOMES:
Incidence of surgical site infections at the midline site (wound) and at the stoma site (wound) that occur within the period from surgery through postop day 42. | 42 Days
  No evidence of infection
Median time to greater than 50% surgical stoma site (wound) closure relative to the stoma site (wound) size at enrollment. | 42 Days
  Median days to greater than 50% closure of the original wound
Area under the plasma concentration versus time curve (AUC) of NM-IL-12 | 1 week
  Area under the plasma concentration versus time curve (AUC) of NM-IL-12
Peak Plasma Concentration (Cmax) of NM-IL-12 | 1 week
  Peak Plasma Concentration (Cmax) of NM-IL-12
Immunogenicity of HemaMax (anti-NM-IL-12 antibodies as a measure of immunogenicity) | 3 months
  anti-NM-IL-12 antibodies as a measure of immunogenicity
Pharmacodynamics of NM-IL-12, Peak Plasma Concentration (Cmax) of IFN-g | 1 week
  Peak Plasma Concentration (Cmax) of IFN-g
Pharmacodynamics of NM-IL-12, Area under the plasma concentration versus time curve (AUC) of IFN-g | 1 week
  Area under the plasma concentration versus time curve (AUC) of IFN-g
Pharmacodynamics of NM-IL-12, Area under the plasma concentration versus time curve (AUC) of IP-10 | 1 week
  Area under the plasma concentration versus time curve (AUC) of IP-10
Pharmacodynamics of NM-IL-12, Peak Plasma Concentration (Cmax) of IP-10 | 1 week
  Peak Plasma Concentration (Cmax) of IFN-g

CONTACTS AND LOCATIONS:
Overall Officials: Grant V Bochicchio, MD, MPH (GB), Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - University of Maryland, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gokhale MS, Vainstein V, Tom J, Thomas S, Lawrence CE, Gluzman-Poltorak Z, Siebers N, Basile LA. Single low-dose rHuIL-12 safely triggers multilineage hematopoietic and immune-mediated effects. Exp Hematol Oncol. 2014 Apr 11;3(1):11. doi: 10.1186/2162-3619-3-11. PMID 24725395